CLINICAL TRIAL: NCT02048813
Title: A Randomized Phase III Study of Ibrutinib (PCI-32765)-Based Therapy vs Standard Fludarabine, Cyclophosphamide, and Rituximab (FCR) Chemoimmunotherapy in Untreated Younger Patients With Chronic Lymphocytic Leukemia (CLL)
Brief Title: Ibrutinib and Rituximab Compared With Fludarabine Phosphate, Cyclophosphamide, and Rituximab in Treating Patients With Untreated Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-00118; NCI-2014-00118 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); E1912; ECOG-E1912; E1912 (Other: ECOG-ACRIN Cancer Research Group); E1912 (Other: CTEP); R01CA193541 (NIH); U10CA021115 (NIH); U10CA180820 (NIH); U24CA196172 (NIH)
Record Dates: First submitted 2014-01-27; First posted 2014-01-29 (Estimated); Results first posted 2023-08-14 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-10

CONDITIONS: Anemia; Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
MeSH Terms: conditions — Anemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Cyclophosphamide; fludarabine phosphate; ibrutinib; Pharmacogenomic Testing; Rituximab; CT-P10

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (ibrutinib, rituximab) (Experimental): Patients receive ibrutinib PO QD on days 1-28. Beginning cycle 2, patients also receive rituximab IV over 4 hours on days 1 and 2 of cycle 2, and day 1 of cycles 3-7. Treatment repeats every 28 days for 7 cycles in the absence of unacceptable toxicity. In the absence of disease progression, patients may continue ibrutinib PO QD for a maximum of 10 years.
  Interventions: Drug: Ibrutinib; Other: Laboratory Biomarker Analysis; Other: Pharmacogenomic Study; Other: Quality-of-Life Assessment; Biological: Rituximab
- Arm B (rituximab, fludarabine phosphate, cyclophosphamide) (Active Comparator): Patients receive rituximab IV over 4 hours on days 1 and 2 of cycle 1, and day 1 of cycles 2-6. Patients also receive fludarabine phosphate IV over 30 minutes and cyclophosphamide IV over 30 minutes on days 1-3. Treatment repeats every 28 days for 6 cycles in the absence of unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Other: Pharmacogenomic Study; Other: Quality-of-Life Assessment; Biological: Rituximab

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
  Arms: Arm B (rituximab, fludarabine phosphate, cyclophosphamide)
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
  Arms: Arm B (rituximab, fludarabine phosphate, cyclophosphamide)
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA 032765; CRA-032765; CRA032765; Imbruvica; PCI 32765; PCI-32765; PCI32765
  Arms: Arm A (ibrutinib, rituximab)
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacogenomic Study — Correlative studies
  Other Names: PHARMACOGENOMIC
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Biological: Rituximab — Given IV
  Other Names: ABP 798; ABP-798; ABP798; BI 695500; BI-695500; BI695500; Blitzima; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT P10; CT-P10; CTP10; GP 2013; GP-2013; GP2013; IDEC 102; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; IDEC102; Ikgdar; Mabtas; MabThera; Monoclonal Antibody IDEC-C2B8; PF 05280586; PF-05280586; PF05280586; Riabni; Ritemvia; Rituxan; Rituximab ABBS; Rituximab ARRX; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar GP2013; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; Rituximab PVVR; Rituximab-abbs; Rituximab-arrx; Rituximab-blit; Rituximab-pvvr; Rituximab-rite; Rituximab-rixa; Rituximab-rixi; Rixathon; Riximyo; RTXM 83; RTXM-83; RTXM83; Ruxience; Truxima

SUMMARY:
This phase III trial studies ibrutinib and rituximab to see how well they work compared to fludarabine phosphate, cyclophosphamide, and rituximab in treating patients with untreated chronic lymphocytic leukemia or small lymphocytic lymphoma. Ibrutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Chemotherapy drugs, such as fludarabine phosphate and cyclophosphamide, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Rituximab is a monoclonal antibody. It binds to a protein called CD20, which is found on B cells (a type of white blood cell) and some types of cancer cells. This may help the immune system kill cancer cells. It is not yet known whether fludarabine phosphate, cyclophosphamide, and rituximab may work better than ibrutinib and rituximab in treating patients with untreated chronic lymphocytic leukemia or small lymphocytic lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the ability of ibrutinib-based induction therapy to prolong progression free survival (PFS) compared to standard fludarabine phosphate, cyclophosphamide, and rituximab (FCR) chemoimmunotherapy for younger patients with chronic lymphocytic leukemia (CLL).

SECONDARY OBJECTIVES:

I. Evaluate overall survival (OS) of patients based on treatment arm. II. Monitor and assess toxicity of treatment with ibrutinib-based induction relative to standard FCR chemotherapy.

III. To compare quality of life (QOL) in CLL patients during the first 6 months of treatment among patients receiving ibrutinib-based induction therapy relative to standard FCR chemoimmunotherapy.

IV. To compare QOL over the long-term in CLL patients receiving continuous therapy using ibrutinib to that of CLL patients who completed FCR therapy.

V. Determine the effect of pretreatment clinical and biological characteristics (e.g. disease stage, immunoglobulin heavy chain variable region gene [IGHV] mutation status, fluorescent in situ hybridization [FISH]) on clinical outcomes (e.g. complete response, PFS) of the different arms.

VI. Determine if the minimal residual disease (MRD) status as assessed by flow cytometry at different time points during and after treatment is an effective surrogate marker for prolonged PFS and overall survival.

VII. Compare the genetic abnormalities and dynamics of intra-clonal architecture of CLL patients before and after treatment with chemoimmunotherapy (CIT) and non-CIT approaches and explore relationships with treatment resistance.

VIII. Explore the effects of FCR and ibrutinib-based therapy on T-cell immune function.

IX. Conduct confirmatory validation genotyping of single nucleotide polymorphisms (SNPs) associated with the efficacy and toxicity of fludarabine-based therapy as in a prior Eastern Cooperative Oncology Group (ECOG) genome-wide association study (GWAS) analysis in the E2997 trial.

X. Evaluate the ability of prognostic model that incorporates clinical and biologic characters to predict a response to therapy and clinical outcome (PFS, OS).

XI. Evaluate signaling networks downstream of the B-cell receptor in patients receiving ibrutinib-based therapy.

XII. Collect relapse samples to study mechanisms of resistance to both FCR and ibrutinib-based therapy.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM A: Patients receive ibrutinib orally (PO) once daily (QD) on days 1-28. Beginning cycle 2, patients also receive rituximab intravenously (IV) over 4 hours on days 1 and 2 of cycle 2, and day 1 of cycles 3-7. Treatment repeats every 28 days for 7 cycles in the absence of unacceptable toxicity. In the absence of disease progression, patients may continue ibrutinib PO QD for a maximum of 10 years.

ARM B: Patients receive rituximab IV over 4 hours on days 1 and 2 of cycle 1, and day 1 of cycles 2-6. Patients also receive fludarabine phosphate IV over 30 minutes and cyclophosphamide IV over 30 minutes on days 1-3. Treatment repeats every 28 days for 6 cycles in the absence of unacceptable toxicity.

After completion of study treatment, patients are followed up for 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CLL according to the National Cancer Institute (NCI)/Internal Workshop on Chronic Lymphocytic Leukemia (IWCLL) criteria or small lymphocytic lymphoma (SLL) according to the World Health Organization (WHO) criteria; this includes previous documentation of:

  * Biopsy-proven small lymphocytic lymphoma or
  * Diagnosis of CLL according to the NCI/IWCLL criteria as evidenced by all of the following:

    * Peripheral blood lymphocyte count of greater than 5 x 10^9/L
    * Immunophenotype consistent with CLL defined as:

      * The predominant population of lymphocytes share both B-cell antigens (cluster of differentiation [CD]19, CD20 [typically dim expression], or CD23) as well as CD5 in the absence of other pan-T-cell markers (CD3, CD2, etc)
      * Clonality as evidenced by kappa or lambda light chain restriction (typically dim immunoglobulin expression)
  * Negative FISH analysis for t(11;14)(immunoglobulin heavy locus [IgH]/cyclin D1 [CCND1]) on peripheral blood or tissue biopsy (e.g. marrow aspirate) or negative immunohistochemical stains for cyclin D1 staining on involved tissue biopsy (e.g. marrow aspirate or lymph node biopsy)
* No prior chemotherapy, Bruton's tyrosine kinase (BTK) inhibitor therapy, or monoclonal anti-body therapy for treatment of CLL or SLL
* Has met at least one of the following indications for treatment:

  * Evidence of progressive marrow failure as manifested by the development of worsening anemia (hemoglobin [Hg] < 11 g/dl) and/or thrombocytopenia (platelets < 100 x 10^9/L)
  * Symptomatic or progressive lymphadenopathy, splenomegaly, or hepatomegaly
  * One or more of the following disease-related symptoms:

    * Weight loss >= 10% within the previous 6 months
    * Grade 2 or 3 fatigue attributed to CLL
    * Fevers > 100.5 Fahrenheit (F) for 2 weeks without evidence of infection
    * Clinically significant night sweats without evidence of infection
  * Progressive lymphocytosis (not due to the effects of corticosteroids) with an increase of > 50% over a two-month period or an anticipated doubling time of less than six months
* Age ≥ 18 years and ≤ 70
* ECOG performance status between 0-2
* Life expectancy of >= 12 months
* Ability to tolerate FCR based therapy
* No deletion of 17p13 on cytogenetic analysis by FISH
* Glomerular filtration rate (GFR) > 40 mL/minute as calculated by the Cockcroft-Gault formula (obtained =< 14 days prior to registration)
* Total bilirubin =< 2.5 x upper limit of normal (ULN) (obtained =< 14 days prior to registration) unless due to Gilbert's disease; for those with a total bilirubin > 2.5 x ULN, a direct bilirubin should be performed and must be < 1.5 mg/dL for Gilbert's to be diagnosed

  * If value is higher due to hepatic involvement by CLL, patient is eligible
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate transaminase [AST])/serum glutamate-pyruvate transaminase (SGPT) (alanine transaminase [ALT]) =< 3.0 x the institutional ULN (obtained =< 14 days prior to registration)

  * If value is higher due to hepatic involvement by CLL, patient is eligible
* Prothrombin time (PT)/international normalized ratio (INR) < 1.5 ULN and partial thromboplastin time (PTT) (activated partial thromboplastin time [aPTT]) < 1.5 X ULN (obtained =< 14 days prior to registration)

  * If value is higher due to hepatic involvement by CLL, patient is eligible
* No active hemolytic anemia requiring immunosuppressive therapy or other pharmacologic treatment; patients who have a positive Coombs test but no evidence of hemolysis are NOT excluded from participation
* No current use of corticosteroids; EXCEPTION: low doses of steroids (< 10 mg of prednisone or equivalent dose of other steroid) used for treatment of non-hematologic medical condition (e.g. chronic adrenal insufficiency) is permitted
* No previous use of corticosteroids for autoimmune complications that have developed since the initial diagnosis of CLL; prior use of corticosteroids for reasons other than treatment of autoimmune complications is allowed
* No other active primary malignancy (other than non-melanomatous skin cancer or carcinoma in situ of the cervix) requiring treatment or limiting expected survival to =< 2 years; NOTE: if there is a history of prior malignancy, they must not be receiving other specific treatment (other than hormonal therapy for their cancer)
* Able to adhere to the study visit schedule and other protocol requirements
* No major surgery within the last 4 weeks (28 days) of first dose of study drug or minor surgery within 3 days of first dose of study drug
* No radiation therapy =< 4 weeks prior to registration
* Patients with human immunodeficiency virus (HIV) infection may be eligible provided they meet the following criteria:

  * CD4-positive cell count >= lower limit of institutional normal
  * HIV viral load < 10,000 copies HIV ribonucleic acid (RNA)/mL (if not on anti-HIV therapy) OR < 50 copies HIV RNA/mL (if on anti-HIV therapy)
  * No evidence of hepatitis B or C infection
  * No evidence of resistant strains of HIV
  * No history of acquired immune deficiency syndrome (AIDS)-defining condition
* Patients must not have any of the following conditions:

  * Congestive heart failure or New York Heart Association Functional Classification III or IV congestive heart failure
  * History of myocardial infarction, unstable angina, or acute coronary syndrome within 6 months prior to registration
  * Recent infections requiring systemic treatment; need to have completed anti-biotic therapy > 14 days before the first dose of study drug
  * Cerebral vascular accident or intracranial bleed within the last 6 months
  * Infection with known chronic, active hepatitis C
  * Serologic status reflecting active hepatitis B or C infection; patients that are positive for hepatitis B core antibody, hepatitis B surface antigen (HBsAg), or hepatitis C antibody must have a negative polymerase chain reaction (PCR) prior to enrollment (PCR positive patients will be excluded)
* Patients are not eligible if they require treatment with a strong cytochrome P450 (CYP) family 3, subfamily A (3A) inhibitor
* Patients may not be on any other investigational agents
* Patients may not have received warfarin or another vitamin K antagonist in the preceding 30 days
* Women must not be pregnant or breast-feeding since this study involves an investigational agent whose genotoxic, mutagenic, and teratogenic effects on the developing fetus and newborn are unknown; female patients of childbearing potential must have a negative serum pregnancy test within 2 weeks prior to registration to rule out pregnancy; female patients who are of non-reproductive potential are those who are post-menopausal by history (i.e. no menses for >= 1 year); OR history of hysterectomy; OR history of bilateral tubal ligation; OR history of bilateral oophorectomy)
* Women of childbearing potential and sexually active males must be strongly advised to use an accepted and effective method of contraception or to abstain from sexual intercourse for 90 days after the last dose of study drug
* Patient must be able to swallow capsules and not have the following conditions:

  * Disease significantly affecting gastrointestinal function
  * Resection of the stomach or small bowel
  * Symptomatic inflammatory bowel disease
  * Ulcerative colitis
  * Partial or complete bowel obstruction
* Patient must not be on any other systemic immunosuppressant therapy other than corticosteroids within 28 days of the first dose of study drug
* Patient must not be vaccinated with live, attenuated vaccines within 4 weeks of first dose of study drug
* Patient must not have any known bleeding disorders (e.g., von Willebrand's disease) or hemophilia
* Patient must not have currently active, clinically significant hepatic impairment (>= moderate hepatic impairment according to the NCI/Child Pugh)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 529 (Actual)
Dates: Start 2014-03-10 (Actual); Primary Completion 2018-10-24 (Actual); Study Completion 2026-10-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Tait D Shanafelt, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (783):
- United States (783):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Regional Hospital, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - PCR Oncology, Arroyo Grande, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Adventist Health Cancer Care Center Chico, Chico, California
  - John Muir Medical Center-Concord, Concord, California
  - Sutter Davis Hospital, Davis, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Marin Cancer Care Inc, Greenbrae, California
  - Marin General Hospital, Greenbrae, California
  - Kaiser Permanente South Bay, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles, Los Angeles, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - Kaiser Permanente-Oakland, Oakland, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente Sacramento Medical Center, Sacramento, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Stanford Cancer Center South Bay, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - John Muir Medical Center-Walnut Creek, Walnut Creek, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - National Jewish Health-Main Campus, Denver, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western States Cancer Research NCORP, Denver, Colorado
  - CommonSpirit Cancer Center Mercy, Durango, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Kaiser Permanente-Lone Tree, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Middlesex Hospital, Middletown, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital-Orange Care Center, Orange, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Lakeland Regional Health Hollis Cancer Center, Lakeland, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Atrium Health Navicent, Macon, Georgia
  - Central Georgia Gynecologic Oncology, Macon, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Rush-Copley Medical Center, Aurora, Illinois
  - OSF Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Ascension Alexian Brothers - Elk Grove Village, Elk Grove Village, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - Hematology Oncology Associates of Illinois-Highland Park, Highland Park, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Duly Health and Care Joliet, Joliet, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Trinity Medical Center, Moline, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Illinois Cancer Specialists-Niles, Niles, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - UW Health Carbone Cancer Center Rockford, Rockford, Illinois
  - Hematology Oncology Associates of Illinois - Skokie, Skokie, Illinois
  - North Shore Medical Center, Skokie, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Ascension Saint Vincent Anderson, Anderson, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Mercy Medical Center - North Iowa, Mason City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Abben Cancer Center, Spencer, Iowa
  - MercyOne Waterloo Cancer Center, Waterloo, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Kansas Institute of Medicine Cancer and Blood Center, Lenexa, Kansas
  - Minimally Invasive Surgery Hospital, Lenexa, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Ochsner Medical Center Kenner, Kenner, Louisiana
  - Ochsner LSU Health Monroe Medical Center, Monroe, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - CHRISTUS Highland Medical Center, Shreveport, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Saint Agnes Hospital, Baltimore, Maryland
  - Beverly Hospital, Beverly, Massachusetts
  - Tufts Medical Center, Boston, Massachusetts
  - Eastern Cooperative Oncology Group, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Beth Israel Deaconess Medical Center/Winchester Center for Cancer Care, Winchester, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Corewell Health Farmington Hills Hospital, Farmington Hills, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - William Beaumont Hospital-Grosse Pointe, Grosse Pointe, Michigan
  - Allegiance Health, Jackson, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Monroe Cancer Center, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Henry Ford Health Providence Novi Hospital, Novi, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Michigan Cancer Specialists, Roseville, Michigan
  - Oakland Colon Rectal Associates, Royal Oak, Michigan
  - Cancer Care Associates PC, Royal Oak, Michigan
  - Comprehensive Medical Center PLLC, Royal Oak, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - Hematology Oncology Consultants PC-Royal Oak, Royal Oak, Michigan
  - Oakland Medical Group, Royal Oak, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Henry Ford Health Providence Southfield Hospital, Southfield, Michigan
  - Premier Hematology Oncology Care, Sterling Heights, Michigan
  - Mitchell Folbe MD PC, Sterling Heights, Michigan
  - Michigan Institute of Urology-Town Center, Troy, Michigan
  - Claudia BR Herke MD PC, Troy, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Hematology Oncology Consultants PC-Troy, Troy, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - Fred and Pamela Buffett Cancer Center - Kearney, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Hematology and Oncology, Lincoln, Nebraska
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Cancer Partners of Nebraska, Lincoln, Nebraska
  - Faith Regional Health Services Carson Cancer Center, Norfolk, Nebraska
  - Great Plains Health Callahan Cancer Center, North Platte, Nebraska
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Nebraska Cancer Specialists - Omaha, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Oncology Hematology West PC, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Regional West Medical Center Cancer Center, Scottsbluff, Nebraska
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Oncology Las Vegas - Henderson, Henderson, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Oncology Las Vegas - Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Wentworth-Douglass Hospital, Dover, New Hampshire
  - Veterans Adminstration New Jersey Health Care System, East Orange, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New York Oncology Hematology PC - Albany Medical Center, Albany, New York
  - Hematology Oncology Associates of Central New York-Auburn, Auburn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Hematology Oncology Associates of CNY at Camillus, Camillus, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - Hematology Oncology Associates of Central New York-Liverpool, Liverpool, New York
  - North Shore University Hospital, Manhasset, New York
  - Garnet Health Medical Center, Middletown, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - University of Rochester, Rochester, New York
  - Hematology Oncology Associates of Central New York-Rome, Rome, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Mission Hospital, Asheville, North Carolina
  - AdventHealth Infusion Center Asheville, Asheville, North Carolina
  - Messino Cancer Centers, Asheville, North Carolina
  - Sampson Radiation Oncology, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - AdventHealth Hendersonville, Hendersonville, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - ECU Health Oncology Kinston, Kinston, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Cleveland Clinic Akron General, Akron, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Geauga Hospital, Chardon, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Oncology Hematology Care Inc-Eden Park, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Dayton Veterans Affairs Medical Center, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lancaster Radiation Oncology, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - UH Seidman Cancer Center at Landerbrook Health Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - Dayton Physicians LLC-Signal Point, Middletown, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Dayton Physicians LLC-Wilson, Sidney, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Mercy Health - Saint Vincent Hospital, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Dayton Physicians LLC - Troy, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University Hospitals Sharon Health Center, Wadsworth, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - UH Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - UPMC Hillman Cancer Center in Coraopolis, Moon Township, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Drexel University School of Medicine, Philadelphia, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC-Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC Jefferson Regional Radiation Oncology, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - Pottstown Hospital, Pottstown, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Hematology and Oncology Associates of North East Pennsylvania, Scranton, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - UPMC Uniontown Hospital Radiation Oncology, Uniontown, Pennsylvania
  - UPMC Washington Hospital Radiation Oncology, Washington, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - UPMC Susquehanna, Williamsport, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - SMC Center for Hematology Oncology Union, Union, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Bristol Regional Medical Center, Bristol, Tennessee
  - Memorial Hospital, Chattanooga, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Wellmont Medical Associates Oncology and Hematology-Johnson City, Johnson City, Tennessee
  - Ballad Health Cancer Care - Kingsport, Kingsport, Tennessee
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Covenant Medical Center-Lakeside, Lubbock, Texas
  - University Hospital, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Danville Regional Medical Center, Danville, Virginia
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - Hematology Oncology Associates of Fredericksburg Inc, Fredericksburg, Virginia
  - Centra Alan B Pearson Regional Cancer Center, Lynchburg, Virginia
  - Sovah Health Martinsville, Martinsville, Virginia
  - Ballad Health Cancer Care - Norton, Norton, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Virginia Mason Bainbridge Island Medical Center, Bainbridge Island, Washington
  - Overlake Medical Center, Bellevue, Washington
  - Swedish Cancer Institute-Eastside Oncology Hematology, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Virginia Mason Federal Way Medical Center, Federal Way, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Tacoma/Valley Radiation Oncology Centers-Gig Harbor, Gig Harbor, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Northwest Cancer Clinic, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Virginia Mason Lynnwood Medical Center, Lynnwood, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Peninsula Cancer Center, Poulsbo, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Tacoma/Valley Radiation Oncology Centers-Puyallup, Puyallup, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Downtown, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Valley, Spokane Valley, Washington
  - Tacoma/Valley Radiation Oncology Centers-Jackson Hall, Tacoma, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Northwest NCI Community Oncology Research Program, Tacoma, Washington
  - Tacoma/Valley Radiation Oncology Centers-Saint Joe's, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - United Hospital Center, Bridgeport, West Virginia
  - WVUH-Berkely Medical Center, Martinsburg, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - HSHS Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Bellin Memorial Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Mercyhealth Hospital and Cancer Center - Janesville, Janesville, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield Medical Center - Ladysmith, Ladysmith, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Waukesha, Waukesha, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Big Horn Basin Cancer Center, Cody, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Derived] O'Connell NS, Zhao F, Lee JW, Ip EH, Peipert JD, Graham N, Smith ML, Gareen IF, Carlos RC, Obeng-Gyasi S, Sparano JA, Shanafelt TD, Thomas ML, Cella D, Wagner LI, Gray R. Importance of Low- and Moderate-Grade Adverse Events in Patients' Treatment Experience and Treatment Discontinuation: An Analysis of the E1912 Trial. J Clin Oncol. 2024 Jan 20;42(3):266-272. doi: 10.1200/JCO.23.00377. Epub 2023 Oct 6. PMID 37801678
- [Derived] Shanafelt TD, Wang XV, Hanson CA, Paietta EM, O'Brien S, Barrientos J, Jelinek DF, Braggio E, Leis JF, Zhang CC, Coutre SE, Barr PM, Cashen AF, Mato AR, Singh AK, Mullane MP, Little RF, Erba H, Stone RM, Litzow M, Tallman M, Kay NE. Long-term outcomes for ibrutinib-rituximab and chemoimmunotherapy in CLL: updated results of the E1912 trial. Blood. 2022 Jul 14;140(2):112-120. doi: 10.1182/blood.2021014960. PMID 35427411
- [Derived] Allan JN, Shanafelt T, Wiestner A, Moreno C, O'Brien SM, Li J, Krigsfeld G, Dean JP, Ahn IE. Long-term efficacy of first-line ibrutinib treatment for chronic lymphocytic leukaemia in patients with TP53 aberrations: a pooled analysis from four clinical trials. Br J Haematol. 2022 Feb;196(4):947-953. doi: 10.1111/bjh.17984. Epub 2021 Dec 5. PMID 34865212
- [Derived] List AF, Sun Z, Verma A, Bennett JM, Komrokji RS, McGraw K, Maciejewski J, Altman JK, Cheema PS, Claxton DF, Luger SM, Mattison RJ, Wassenaar TR, Artz AS, Schiffer CA, Litzow MR, Tallman MS. Lenalidomide-Epoetin Alfa Versus Lenalidomide Monotherapy in Myelodysplastic Syndromes Refractory to Recombinant Erythropoietin. J Clin Oncol. 2021 Mar 20;39(9):1001-1009. doi: 10.1200/JCO.20.01691. Epub 2021 Jan 13. PMID 33439748
- [Derived] Shanafelt TD, Wang XV, Kay NE, Hanson CA, O'Brien S, Barrientos J, Jelinek DF, Braggio E, Leis JF, Zhang CC, Coutre SE, Barr PM, Cashen AF, Mato AR, Singh AK, Mullane MP, Little RF, Erba H, Stone RM, Litzow M, Tallman M. Ibrutinib-Rituximab or Chemoimmunotherapy for Chronic Lymphocytic Leukemia. N Engl J Med. 2019 Aug 1;381(5):432-443. doi: 10.1056/NEJMoa1817073. PMID 31365801

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on January 31, 2014 and closed to accrual on June 9, 2016. A total of 529 patients were enrolled on this study.
Groups:
- Arm A (Ibrutinib, Rituximab): Patients receive ibrutinib 420 mg orally (PO) once daily (QD) on days 1-28. Beginning cycle 2, patients also receive rituximab 50 mg/m2 intravenously (IV) over 4 hours on days 1 and 2 of cycle 2, and rituximab 500 mg/m2day 1 of cycles 3-7. Treatment repeats every 28 days for 7 cycles in the absence of unacceptable toxicity. In the absence of disease progression, patients may continue ibrutinib PO QD.
- Arm B (Rituximab, Fludarabine Phosphate, Cyclophosphamide): Patients receive rituximab IV over 4 hours on days 1 (50 mg/m2) and 2 (325 mg/m2) of cycle 1, and day 1 (500 mg/m2) of cycles 2-6. Patients also receive fludarabine phosphate at 25 mg/m2 IV over 30 minutes and cyclophosphamide at 250 mg/m2 IV over 30 minutes on days 1-3. Treatment repeats every 28 days for 6 cycles in the absence of unacceptable toxicity.
Period: Overall Study
Arm/Group | Arm A (Ibrutinib, Rituximab) | Arm B (Rituximab, Fludarabine Phosphate, Cyclophosphamide)
Started | 354 | 175
Completed | 0 | 105
Not Completed | 354 | 70
Not completed — Still on treatment | 279 | 0
Not completed — Adverse Event | 40 | 38
Not completed — Disease progression | 13 | 3
Not completed — Withdrawal by Subject | 7 | 8
Not completed — Death | 2 | 1
Not completed — Complication | 2 | 2
Not completed — Non-protocol therapy | 0 | 1
Not completed — Second primary cancer | 2 | 0
Not completed — Insurance | 2 | 0
Not completed — Wound infection/healing | 2 | 0
Not completed — Missed appointment | 3 | 0
Not completed — Never started treatment | 2 | 17

BASELINE CHARACTERISTICS:
Population: All randomized patients were included in this analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Ibrutinib, Rituximab) | Arm B (Rituximab, Fludarabine Phosphate, Cyclophosphamide) | Total
Number analyzed (Participants) | 354 | 175 | 529
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.7 (7.5) | 56.7 (7.2) | 56.7 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118 | 55 | 173
  Male | 236 | 120 | 356
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 3 | 10
  Not Hispanic or Latino | 333 | 167 | 500
  Unknown or Not Reported | 14 | 5 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 5 | 3 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 23 | 6 | 29
  White | 318 | 160 | 478
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 8 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) Rate at 3 Years
Description: PFS was defined as the time from randomization to CLL progression or death, whichever occurred first. Progression is characterized by any of the following:
  * ≥ 50% increase from nadir since start of treatment (tx) in the sum of the products of at least 2 lymph nodes on 2 consecutive examinations 2 weeks apart
  * ≥ 50% increase from nadir since start of tx in the size of liver and/or spleen
  * ≥ 50% increase in the absolute number of circulating lymphocytes not due to tumor flare reaction. The absolute lymphocyte count must be ≥ 5x10^9/L to qualify as disease progression.
  * Transformation to a more aggressive histology (e.g. Richter's syndrome or prolymphocytic leukemia with > 55% prolymphocytes). For patients who achieve a complete response or nodular partial response, progression is defined as recurrence of circulating leukemia cell clone in the peripheral blood and an absolute lymphocyte count > 5x10^9/L and/or recurrence of palpable lymphadenopathy > 1.5 cm by physical exam.
Time Frame: Assessed every 3 months until progression up to 4 years and 8 months
Population: All randomized patients were included in this analysis.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Arm A (Ibrutinib, Rituximab) | Arm B (Rituximab, Fludarabine Phosphate, Cyclophosphamide)
Number analyzed (Participants) | 354 | 175
Proportion of participants | 0.894 [0.86 to 0.93] | 0.729 [0.653 to 0.813]
Statistical Analysis 1: Comparison: Arm A (Ibrutinib, Rituximab) vs Arm B (Rituximab, Fludarabine Phosphate, Cyclophosphamide); Test type: Superiority; p < .001, Log Rank; Hazard Ratio (HR) = 0.35, 95% CI 2-sided [0.22 to 0.56]

2. Secondary Outcome: Overall Survival (OS) Rate at 3 Years
Description: Overall survival was defined as time from randomization to death from any cause or date last known alive. Overall survival rate at 3 years was estimated using the method of Kaplan-Meier.
Time Frame: Assessed every 3 months until progression; after progression, assessed every 3 months for first 2 years, every 6 months for years 3-5, up to 4 years and 8 months
Population: All randomized patients were included in this analysis.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Arm A (Ibrutinib, Rituximab) | Arm B (Rituximab, Fludarabine Phosphate, Cyclophosphamide)
Number analyzed (Participants) | 354 | 175
Proportion of participants | 0.988 [0.976 to 1.00] | 0.915 [0.862 to 0.970]
Statistical Analysis 1: Comparison: Arm A (Ibrutinib, Rituximab) vs Arm B (Rituximab, Fludarabine Phosphate, Cyclophosphamide); Test type: Superiority; p < .001, Log Rank; Hazard Ratio (HR) = 0.17, 95% CI 2-sided [0.05 to 0.54]

3. Secondary Outcome: The Functional Assessment of Cancer Therapy - Leukemia (FACT-Leu) Trial Outcome Index (TOI) Score at 6 Months
Description: The Functional Assessment of Cancer Therapy - Leukemia (FACT-Leu) Trial Outcome Index (TOI) is comprised of the physical well-being (PWB) and functional well-being (FWB) components of the FACT-General (FACT-G) and the leukemia subscale. The FACT-Leu TOI contains a total of 31 items, with scores ranging from 0 to 124. The higher the score, the better the quality of life (QOL).
Time Frame: Assessed at 6 months
Reporting Status: Not Posted

4. Secondary Outcome: The Functional Assessment of Cancer Therapy - Leukemia (FACT-Leu) Trial Outcome Index (TOI) Score at 12 Months
Description: as for outcome 3
Time Frame: Assessed at 12 months
Reporting Status: Not Posted

5. Secondary Outcome: The Association Between Baseline Rai Stage and Complete Response (CR) Rate
Description: Patients are classified as stage 0-IV according to the Rai system and categorized into one of the three risk groups:
  Low risk - Stage 0 Intermediate risk - Stage I or II High risk - Stage III or IV
  CR requires all of the following for at least 2 months:
  * Absence of lymphadenopathy by physical examination on 2 occasions at least 4 weeks apart and appropriate radiographic techniques. For patients whose only measurable disease at the time of enrollment is on CT scan, a CT scan is required and all lymph nodes must be ≤ 1.5 cm before classifying the patient a CR.
  * Absence of hepatomegaly or splenomegaly by physical examination
  * Absence of constitutional symptoms due to disease
  * Normal complete blood count
  * One marrow aspirate and biopsy should be performed 52 weeks after Day 1 of cycle 1 among patients with clinical and laboratory evidence of a CR to document a CR. The marrow sample must be at least normocellular with < 30% of nucleated cells being lymphocytes.
Time Frame: Assessed at baseline, every 3 months for the first 2 years, and every 6 months for years 3-5
Reporting Status: Not Posted

6. Secondary Outcome: Progression-free Survival (PFS) by Measurable Residual Disease (MDR) Status at 2 Years
Description: PFS was defined as time from randomization to progression or death. Progression is characterized by any of the following:
  * ≥ 50% increase from nadir since start of treatment (tx) in the sum of the products of ≥ 2 lymph nodes on 2 consecutive exams 2 weeks apart
  * ≥ 50% increase from nadir since start of tx in the size of liver and/or spleen
  * ≥ 50% increase in the absolute number of circulating lymphocytes not due to tumor flare reaction. The absolute lymphocyte count must be ≥ 5x10^9/L to qualify as progression.
  * Transformation to a more aggressive histology. For patients with a complete response or nodular partial response, progression is defined as recurrence of circulating leukemia cell clone in the peripheral blood and an absolute lymphocyte count > 5x10^9/L and/or recurrence of palpable lymphadenopathy >1.5 cm by physical exam.
  MRD status was evaluated at 2 years and samples with <=20 monotypic events or an MRD level of <10^-4 were classified as undetectable MRD.
Time Frame: Assessed every 3 months until progression up to 5 years
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Distribution of Genetic Abnormalities Before and After Treatment
Description: Genetic abnormalities are assessed at baseline and longitudinally during treatment as well as after treatment. Distribution of genetic abnormalities are reported.
Time Frame: Assessed at baseline, and 3, 6, 12, 15, 18, 24, 36 months
Reporting Status: Not Posted

8. Other Pre Specified Outcome: T-cell Counts at 12 Months
Description: T-cell counts will be measured at 12 months.
Time Frame: Assessed at 12 months
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Association Between Single Nucleotide Polymorphisms (SNPs) and PFS
Description: PFS was defined as time from randomization to progression or death, whichever occurred first. Progression is characterized by any of the following:
  * ≥ 50% increase from nadir since start of treatment (tx) in the sum of the products of ≥2 lymph nodes on 2 consecutive examinations 2 weeks apart
  * ≥ 50% increase from nadir since start of tx in the size of liver and/or spleen
  * ≥ 50% increase in the absolute number of circulating lymphocytes not due to tumor flare reaction. The absolute lymphocyte count must be ≥ 5x10^9/L to qualify as progression.
  * Transformation to a more aggressive histology. For patients who achieve a complete response or nodular partial response, progression is defined as recurrence of circulating leukemia cell clone in the peripheral blood and an absolute lymphocyte count > 5x10^9/L and/or recurrence of palpable lymphadenopathy > 1.5 cm by physical exam.
  The distribution of PFS by SNPs will be reported.
Time Frame: Assessed every 3 months until progression; after progression, assessed every 3 months for first 2 years, every 6 months for years 3-5
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Prognostic Model to Predict PFS
Description: A prognostic model that incorporates clinical and biologic characters to predict PFS will be developed.
Time Frame: as for outcome 9
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Signaling Networks Downstream of the B-cell Receptor
Description: Evaluation of signaling networks downstream of the B-cell receptor in patients receiving Ibrutinib-based therapy.
Time Frame: Assessed at baseline and 3, 6, 12, 15, 18, 24, 36 months
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Collection of Relapse Samples
Description: Collection of relapse samples to study mechanisms of resistance to protocol treatments.
Time Frame: Assessed at relapse
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Assessed every 4 weeks while on treatment and for 30 days after the end of treatment, up to 4.5 years
Description: Only patients who started protocol therapy are included in the analysis of adverse events. All registered patients are included in the analysis of all-cause mortality.
Arm/Group | Arm A (Ibrutinib, Rituximab) | Arm B (Rituximab, Fludarabine Phosphate, Cyclophosphamide)
All-Cause Mortality (participants affected / at risk) | 4/354 | 10/175
Serious Adverse Events (participants affected / at risk) | 270/352 | 132/158
Other Adverse Events (participants affected / at risk) | 348/352 | 154/158
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Ibrutinib, Rituximab) (N=352) | Arm B (Rituximab, Fludarabine Phosphate, Cyclophosphamide) (N=158)
Ear pain (Ear and labyrinth disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 16 | 25
Febrile neutropenia (Blood and lymphatic system disorders) | 8 | 25
Hemolysis (Blood and lymphatic system disorders) | 0 | 4
Leukocytosis (Blood and lymphatic system disorders) | 36 | 1
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 | 1
Asystole (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 20 | 0
Atrial flutter (Cardiac disorders) | 3 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 5 | 0
Chest pain - cardiac (Cardiac disorders) | 2 | 0
Conduction disorder (Cardiac disorders) | 1 | 0
Heart failure (Cardiac disorders) | 3 | 0
Pericardial effusion (Cardiac disorders) | 2 | 0
Pericardial tamponade (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 2 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Chills (General disorders) | 1 | 1
Edema limbs (General disorders) | 1 | 0
Fatigue (General disorders) | 8 | 4
Fever (General disorders) | 2 | 2
Infusion related reaction (General disorders) | 1 | 1
Multi-organ failure (General disorders) | 2 | 0
Pain (General disorders) | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 9 | 3
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 0
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 9 | 1
Gastric hemorrhage (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 3 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Allergic reaction (Immune system disorders) | 1 | 0
Immune system disorders - Other, specify (Immune system disorders) | 2 | 1
Encephalitis infection (Infections and infestations) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 1 | 1
Hepatitis viral (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 22 | 4
Papulopustular rash (Infections and infestations) | 1 | 0
Penile infection (Infections and infestations) | 1 | 0
Scrotal infection (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 7 | 5
Sinusitis (Infections and infestations) | 0 | 2
Skin infection (Infections and infestations) | 5 | 1
Soft tissue infection (Infections and infestations) | 3 | 0
Upper respiratory infection (Infections and infestations) | 3 | 3
Urinary tract infection (Infections and infestations) | 6 | 1
Wound infection (Infections and infestations) | 1 | 0
Infections and infestations - Other, specify (Infections and infestations) | 16 | 1
Intraoperative hemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 8 | 0
Alkaline phosphatase increased (Investigations) | 2 | 0
Aspartate aminotransferase increased (Investigations) | 7 | 0
Blood bilirubin increased (Investigations) | 8 | 0
CD4 lymphocytes decreased (Investigations) | 0 | 1
Creatinine increased (Investigations) | 1 | 0
Ejection fraction decreased (Investigations) | 2 | 0
Lymphocyte count decreased (Investigations) | 25 | 103
Lymphocyte count increased (Investigations) | 97 | 22
Neutrophil count decreased (Investigations) | 102 | 72
Platelet count decreased (Investigations) | 14 | 26
Weight gain (Investigations) | 4 | 0
White blood cell decreased (Investigations) | 23 | 64
Investigations - Other, specify (Investigations) | 3 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 4 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 2
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 4 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0
Tumor lysis syndrome (Metabolism and nutrition disorders) | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal and connective tissue disorder - Other, spe (Musculoskeletal and connective tissue disorders) | 2 | 0
Cognitive disturbance (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0
Encephalopathy (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 4 | 1
Intracranial hemorrhage (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 1
Stroke (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 3 | 0
Leukemia secondary to oncology chemotherapy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 1
Neoplasms benign, malignant and unspecified (incl cysts and (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Depression (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Respiratory, thoracic and mediastinal disorders - Other, spe (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Hematuria (Renal and urinary disorders) | 1 | 0
Renal hemorrhage (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 1
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 2 | 0
Hematoma (Vascular disorders) | 3 | 1
Hypertension (Vascular disorders) | 44 | 3
Hypotension (Vascular disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 0 | 1
Vascular disorders - Other, specify (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Ibrutinib, Rituximab) (N=352) | Arm B (Rituximab, Fludarabine Phosphate, Cyclophosphamide) (N=158)
Anemia (Blood and lymphatic system disorders) | 183 | 99
Atrial fibrillation (Cardiac disorders) | 27 | 0
Palpitations (Cardiac disorders) | 30 | 1
Chills (General disorders) | 20 | 17
Edema limbs (General disorders) | 61 | 14
Fatigue (General disorders) | 235 | 105
Fever (General disorders) | 42 | 32
Infusion related reaction (General disorders) | 28 | 39
Pain (General disorders) | 22 | 3
General disorders and administration site conditions - Other (General disorders) | 26 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 31 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 29 | 8
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 111 | 16
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 65 | 5
Abdominal pain (Gastrointestinal disorders) | 26 | 4
Constipation (Gastrointestinal disorders) | 39 | 38
Diarrhea (Gastrointestinal disorders) | 146 | 24
Dry mouth (Gastrointestinal disorders) | 25 | 3
Dyspepsia (Gastrointestinal disorders) | 34 | 4
Gastroesophageal reflux disease (Gastrointestinal disorders) | 36 | 4
Mucositis oral (Gastrointestinal disorders) | 60 | 12
Nausea (Gastrointestinal disorders) | 117 | 96
Vomiting (Gastrointestinal disorders) | 30 | 40
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 25 | 2
Skin infection (Infections and infestations) | 22 | 1
Upper respiratory infection (Infections and infestations) | 44 | 13
Infections and infestations - Other, specify (Infections and infestations) | 23 | 4
Bruising (Injury, poisoning and procedural complications) | 117 | 3
Alanine aminotransferase increased (Investigations) | 49 | 17
Alkaline phosphatase increased (Investigations) | 37 | 20
Aspartate aminotransferase increased (Investigations) | 61 | 27
Blood bilirubin increased (Investigations) | 70 | 22
Creatinine increased (Investigations) | 74 | 14
Lymphocyte count decreased (Investigations) | 80 | 80
Lymphocyte count increased (Investigations) | 132 | 12
Neutrophil count decreased (Investigations) | 117 | 80
Platelet count decreased (Investigations) | 181 | 104
Weight gain (Investigations) | 25 | 4
White blood cell decreased (Investigations) | 74 | 108
Anorexia (Metabolism and nutrition disorders) | 39 | 28
Hyperglycemia (Metabolism and nutrition disorders) | 31 | 9
Hyperkalemia (Metabolism and nutrition disorders) | 21 | 4
Hyperuricemia (Metabolism and nutrition disorders) | 41 | 6
Hypoalbuminemia (Metabolism and nutrition disorders) | 21 | 4
Hypocalcemia (Metabolism and nutrition disorders) | 42 | 18
Hypokalemia (Metabolism and nutrition disorders) | 19 | 6
Hypophosphatemia (Metabolism and nutrition disorders) | 9 | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 108 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 19 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 112 | 20
Pain in extremity (Musculoskeletal and connective tissue disorders) | 25 | 2
Musculoskeletal and connective tissue disorder - Other, spe (Musculoskeletal and connective tissue disorders) | 42 | 2
Dizziness (Nervous system disorders) | 44 | 15
Dysgeusia (Nervous system disorders) | 19 | 9
Headache (Nervous system disorders) | 89 | 25
Peripheral sensory neuropathy (Nervous system disorders) | 41 | 10
Blurred vision (Eye disorders) | 24 | 3
Anxiety (Psychiatric disorders) | 12 | 8
Insomnia (Psychiatric disorders) | 27 | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 36 | 11
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 32 | 18
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 27 | 1
Hematuria (Renal and urinary disorders) | 29 | 2
Urinary frequency (Renal and urinary disorders) | 1 | 9
Hypertension (Vascular disorders) | 105 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-20): https://cdn.clinicaltrials.gov/large-docs/13/NCT02048813/Prot_SAP_000.pdf